CLINICAL TRIAL: NCT05354232
Title: Home-based Transcranial Direct Current Stimulation (tDCS) for Treatment of Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, Division Chief - Neuropsychiatry & Neuromodulation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P000362
Record Dates: First submitted 2022-04-07; First posted 2022-04-29 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Attention Deficit Disorder; Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized during the first study visit to the 2mA, 1mA, or sham conditions. Subjects will not change dose throughout study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Soterix devices allow for effective and automated double-blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- 2mA transcranial direct current stimulation (Experimental)
  Interventions: Device: 2 mA transcranial direct current stimulation (tDCS)
- 1mA transcranial direct current stimulation (Experimental)
  Interventions: Device: 1 mA transcranial direct current stimulation (tDCS)
- Sham transcranial direct current stimulation (Sham Comparator)
  Interventions: Device: Sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: 2 mA transcranial direct current stimulation (tDCS) — tDCS is a non-invasive neuromodulatory technique that has previously demonstrated the ability to transiently modulate cognitive domains in both healthy and psychiatric populations. In the 2mA condition, the investigators will assist the administration of a 2mA current stimulation from the device.
  Arms: 2mA transcranial direct current stimulation
Device: 1 mA transcranial direct current stimulation (tDCS) — tDCS is a non-invasive neuromodulatory technique that has previously demonstrated the ability to transiently modulate cognitive domains in both healthy and psychiatric populations. In the 1mA condition, the investigators will assist the administration of a 1mA current stimulation from the device.
  Arms: 1mA transcranial direct current stimulation
Device: Sham transcranial direct current stimulation (tDCS) — tDCS is a non-invasive neuromodulatory technique that has previously demonstrated the ability to transiently modulate cognitive domains in both healthy and psychiatric populations. In the sham condition, the investigators will assist the administration of a sham stimulation from the device.
  Arms: Sham transcranial direct current stimulation

SUMMARY:
The investigators are investigating whether home-based tDCS over the course of four weeks can improve ADHD symptom severity and improve dysexecutive functioning (cognitive control). Further, the investigators are investigating whether there is a dose-dependent response to tDCS.

DETAILED DESCRIPTION:
This mechanistic clinical trial will be the first of its kind to assess the clinical and cognitive efficacy of tDCS, and its relationship to physiological target engagement. It will also provide critical knowledge about tDCS dosing in a therapeutic context (i.e. 30 days of daily tDCS). Last, it will assess the feasibility and acceptability of home-based neuromodulation therapies for ADHD, reducing the most significant obstacle for the implementation of devices therapies (i.e. daily visits to the hospital for several weeks) and facilitating access to advanced therapeutics to a large population of patients with ADHD. An additional goal of the proposed study is to assess the feasibility and acceptability of home-based neuromodulation therapies for ADHD, reducing the most significant obstacle for the implementation of devices therapies (i.e. daily visits to the hospital for several weeks) and facilitating access to advanced therapeutics to a large population of patients with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients 18-65 years of age
2. A diagnosis of ADD/ADHD or meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.

Exclusion Criteria:

1. Contraindication to tDCS: history or epilepsy, metallic implants in the head and neck, brain stimulators, vagus nerve stimulators, VP shunt, pacemakers, pregnancy.
2. Active substance dependence (except for tobacco).
3. Pregnant or nursing females.
4. Inability to participate in testing procedures.
5. Premorbid neurological conditions (including neurovascular and neurodegenerative diseases such as traumatic brain injury, stroke, Parkinson's, AD and other dementias) and severe psychiatric disorders (bipolar disorder, schizophrenia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
P300 Amplitude during Erickson Flanker Task | Week 1 - Week 8 of Study
  P300, an electrophysiological feature theorized to represent executive functioning, has been previously shown to be notably diminished during the Erickson Flanker Task (EFT) . We will be administering this task to assess changes in P300 during the EFT, and if any changes are related to subjects' assigned condition.
Global Assessment of Functioning (GAF) Scale | Week 1 - Week 8 of Study
  investigators will use GAF scale to assess the potential feasibility of at-home tDCS for future research.
Adult ADHD Self-Report Scale | Week 1 - Week 8 of Study
  Investigators will assess changes to these questionnaires in reference to assigned stimulation group to assess changes to ADHD symptomatology across study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Camprodon, MD, PHD, MPH, Principal Investigator — MGB: Division of Neuropsychiatry and Neuromodulation
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD for the current study available to other researchers.

REFERENCES:
- [Background] Zhou AQ. [Report of 20 cases of ventricular septal defects with patent ductus arteriosus in children]. Zhonghua Xin Xue Guan Bing Za Zhi. 1982 Dec;10(4):274-5. No abstract available. Chinese. PMID 7160297